CLINICAL TRIAL: NCT06765356
Title: Pragmatic Evaluation of a Pentaspline Pulsed Field Ablation System to Treat Atrial Fibrillation and Related Arrhythmias
Acronym: PROSPECT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director, Cardiac Arrhythmia Service, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANY 24-02-283
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Long-standing Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; A-Fib; Treatment of Atrial Fibrillation; A-Fib Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Non-randomized, interventional clinical study to determine the safety and efficacy in using Pulse Field Ablation with the FARAPULSE Catheter System in the treatment of persistent or paroxysmal atrial fibrillation. All patients will receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Patients with Atrial Fibrillation (Experimental): All patients will receive treatment using the Farapulse catheter system (Farawave catheter used in combination with the Farastar generator).
  Interventions: Device: Farapulse Catheter System; Drug: Low-dose Colchicine

INTERVENTIONS:
Device: Farapulse Catheter System — The FARAWAVE PFA Catheter is a sterile, single use, over-the-wire, non-deflectable device that is used with the FARASTAR Catheter Connection Cable and FARASTAR Generator to enable delivery of Pulsed Field Ablation energy for irreversible electroporation. The FARAWAVE PFA Catheter has five (5) variably deployable splines. The five splines are undeployed during insertion and removal and during use can deploy continuously from an undeployed state through a partially deployed ("basket-shaped") configuration to a fully deployed ("flower-shaped") configuration with five petals.
Drug: Low-dose Colchicine — For participants in the colchicine sub-study, 0.3 mg BID Colchicine. Colchicine will be prescribed to the patient starting 5 days prior to ablation. Patient will continue the colchicine for 3 weeks post-ablation.

SUMMARY:
The purpose of this pragmatic study is to evaluate the safety, performance and effectiveness of the FARAPULSE catheter system (FARAWAVE catheter used in combination with the FARASTAR generator), to treat patients with atrial fibrillation during clinically-indicated ablation procedures

DETAILED DESCRIPTION:
By virtue of its efficiency, safety profile, and potential for improved efficacy, there is tremendous excitement about the role of pulsed field ablation (PFA) to treat atrial fibrillation. Indeed, multiple FDA IDE clinical trials on PFA have been, or are being, conducted to treat AF. However, most FDA pivotal trials studying PFA enroll very selected populations and have highly focused inclusion/exclusion criteria and, typically only paroxysmal or persistent AF patients with limited upper age criteria are included, failure of Class I/III AADs is often required, and other disease states that may particularly benefit from PFA (e.g., PFA might be particularly effective in treating HCM pts with their thickened atrial tissue).

In observational European studies of the FARAPULSE catheter system, the technology has proved quite safe and effective in treating most patients with AF. It is a highly efficient ablation system, and can be employed with only deep sedation, and without the need for endotracheal intubation. In addition to the FARAWAVE catheter performing PV isolation and ablation of the posterior left atrium, in the MANIFEST-PF post-approval study of EU experience, the FARAWAVE catheter has also been shown able to create other relevant ablation lesions such as cavo-tricuspid isthmus ablation for typical atrial flutter, or a mitral isthmus line for mitral isthmus flutter.

The FARAWAVE multielectrode pentaspline PFA catheter is the study device. It can be deployed in a basket or flower configuration: 1) Both configurations can be used to isolate PVs, 2) The flower configuration can be used to ablate the posterior wall, and 3) Flower configuration for creation of CTI or Mitral Isthmus Lines.

The ablation procedure will typically follow the below sequence:

* Pulmonary Vein Isolation (PVI) to be achieved in all patients with atrial fibrillation
* Posterior wall Ablation: will be used in all persistent/LS-Per AF patients, and as per operator discretion, some paroxysmal AF patients
* Additional ablation lesion sets are per investigators' discretion:

  * Cavo-tricuspid isthmus line
  * Mitral Isthmus Line
  * Regional fractionation clusters (allowed but not encouraged)
  * Any micro-/macro-reentrant atrial tachycardia's
* When PFA is performed next to a coronary artery (eg, CTI or mitral isthmus lines), a nitroglycerin pretreatment protocol will be employed as per study protocol.
* As part of the ablation procedure, any safety assessments that are considered important (e.g., EGD, coronary angiography, etc.) may be performed as per the investigators' discretion; these data will also be collected.
* For a lesion set that cannot be performed using the FARAPULSE catheter technology, a conventional FDA-approved ablation catheter may be used to complete the procedure as per whatever is optimal for the patient outcome

This study is a prospective, multi-center, non-randomized, investigator-initiated IDE clinical study to determine the safety and efficacy of the recently FDA-approved FARAPULSE system to treat the "usual" patients presenting in clinical practice for catheter ablation of AF. (An IDE is required because the approval for the FARAPULSE system: i) only includes paroxysmal AF patients, and ii) doesn't include the technology's use for linear lesions such as the cavo-tricuspid isthmus line. Participants will be followed for 12-months post-procedure.

There is an optional randomized sub-study looking at the utility of peri-procedural low-dose colchicine in attenuating PFA-related pericardial inflammation and its negative effects (symptoms and atrial arrhythmias). Participants will start low-dose colchicine 5 days prior to PFA procedure and continue up to 3 weeks post-PFA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with atrial fibrillation with or without concomitant atrial flutter by ECG at some point in the past, and by any criteria (ECG or clear symptoms within the past year)

  * Previous catheter ablation for other arrhythmias (including left-sided ablation, but not for AF) is allowed
* Planned for a clinically-indicated catheter ablation procedure for managing paroxysmal or persistent atrial fibrillation in accordance with the following recommendations in the ACC/AHA/ACCP/HRS guidelines

  * In patients with symptomatic AF in whom antiarrhythmic drugs have been ineffective, contraindicated, not tolerated or not preferred, and continued rhythm control is desired, catheter ablation is useful to improve symptoms.(Class 1)
  * In selected patients (generally younger with few comorbidities) with symptomatic paroxysmal AF in whom rhythm control is desired, catheter ablation is useful as first-line therapy to improve symptoms and reduce progression to persistent AF. (Class 1)
  * In patients (other than younger with few comorbidities) with symptomatic paroxysmal or persistent AF who are being managed with a rhythm-control strategy, catheter ablation as first-line therapy can be useful to improve symptoms. (Class 2a)
  * In selected patients with asymptomatic or minimally symptomatic AF, catheter ablation may be useful for reducing progression of AF and its associated complications. (Class 2b)
  * In patients who present with a new diagnosis of HFrEF and AF, arrhythmia-induced cardiomyopathy should be suspected, and an early and aggressive approach to AF rhythm control is recommended. (Class 1)
  * In appropriate patients with AF and HFrEF who are on GDMT, and with reasonable expectation of procedural benefit, catheter ablation is beneficial to improve symptoms, QOL, ventricular function, and cardiovascular outcomes. (Class 1)
  * In appropriate patients with symptomatic AF and HFpEF with reasonable expectation of benefit, catheter ablation can be useful to improve symptoms and improve QOL. (Class 2a)
  * In athletes who develop AF, catheter ablation with PVI is a reasonable strategy for rhythm control because of its effectiveness and low risk of detrimental effect on exercise capacity. (Class 2a)
* Have in place or have plans for implantation of a loop recorder, pacemaker or cardiac defibrillator capable of recording atrial rhythm (e.g. dual chamber) (ideally, this implantable device would be present for at least 4 weeks pre-PFA)
* Able and willing to provide written consent and comply with all testing and follow-up requirements

Exclusion Criteria:

* Documented "active" left atrial thrombus (patients may later undergo the procedure if this is no longer present, eg, with anticoagulation treatment)
* Reversible cause of AF (e.g., post-operative, thyroid disorder, etc.)
* Conditions that make an AF ablation procedure unlikely to be successful (e.g., advanced infiltrative cardiomyopathies like amyloid, severe mitral stenosis or regurgitation, and cor pulmonale)
* PCI/STEMI within the prior 1 month
* Active systemic infection or sepsis
* Contraindication to all anticoagulation
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude an ablation procedure
* Women who are pregnant, lactating, or who are of childbearing age and plan on becoming pregnant during this trial.
* Life expectancy or other disease processes likely to limit survival to less than 12 months
* Currently, enrolled in an investigational study evaluating another device, biologic, or drug, that would interfere with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Acute Procedural Success | at the end of the procedure (approximately 60 minutes)
  Acute Procedural Success is defined as confirmation of entrance block in all targeted PVs, and acute block of all linear lesions that are attempted (eg, CTI or mitral isthmus line). (The use of a non-study catheter for PVI will be considered an effectiveness failure; however, use of a non-study catheter for ablation unrelated to PVI will be noted, but not considered a treatment failure)

SECONDARY OUTCOMES:
Number of Chronic Single-Procedure Success | up to 12 months post procedure
  Chronic Single-Procedure Success is defined as freedom from all of the following:
  * Any Detectable AF, AFL or AT;
  * Any re-ablation for AF, AFL or AT;
  * Any cardioversion for AF, AFL or AT;
  * Any use of a non-Failed Class I/III AAD or Amiodarone
  Where "Detectable AF, AFL or AT" refers to either of the following as recorded by the ICM:
  * Symptomatic (patient-initiated) recording containing ≥ 30 seconds of continuous AF or AT/AFL
  * Automatically-detected AF or AT/AFL episodes measured at ≥1 hour in duration (asymptomatic)
Number of Participant to Achieve Linear Lesion Bidirectional Block | at the end of the procedure (approximately 60 minutes)
  Ability to achieve linear lesion bidirectional block using the Farawave catheter alone; for this endpoint, all linear lesions (CTI and Mitral Isthmus) will be aggregated. This will be ascertained acutely after either a 20 min waiting period or despite pharmacologic stress (eg., IV adenosine or IV isoproterenol).
Incidence of Primary Adverse Events (PAEs) | within 7 days of procedure
  Incidence of Primary Adverse Events (PAEs) (within 7 days of the initial procedure). PAEs include the following AEs:
  * Atrio-Esophageal Fistula
  * Phrenic Nerve Paralysis
  * Cardiac Tamponade/perforation
  * Pulmonary Vein Stenosis
  * Death
  * Stroke/CVA
  * Major Vascular Access
  * Complication/Bleeding
  * Thromboembolism
  * Myocardial Infarction TIA
  * Device or procedure related death
  * pulmonary vein stenosis and atrio-esophageal fistula that occur greater than one week (7 days) post-procedure are also considered and analyzed as primary AEs.
Number of patients who developed pericarditis | within 2 weeks from procedure, and at 7 days follow-up visit
  Number of patients who developed clinical pericarditis within 2 weeks following ablation. This will be ascertained by comprehensive chart review plus at the routine post-ablation follow-up phone visit at 7 days
Incidence of Serious Adverse Device Effects (SADEs) | end of study at 12 months
  Incidence of Serious Adverse Device Effects (SADEs)
Incidence of Gastrointestinal symptoms | end of study at 12 months
  Incidence of Gastrointestinal symptoms (necessitating cessation of colchicine therapy) for participants in the substudy
Freedom from detectable AF, AFL or AT off AADs | end of study 12 months
  Freedom from detectable AF, AFL or AT off AADs, defining detectable AF, AFL or AT as Freedom from detectable AF, AFL or AT
Number of patients who achieve CT isthmus block | end of study 12 months
  Number of patients achieving CT isthmus block using the Farawave catheter alone will be recorded.
Freedom from persistent AF at 12 months off AADs | end of study 12 months
  Freedom from persistent AF at 12 months off AADs
Freedom from symptomatic AT/AF/AFL recurrence | end of study 12 months
  Freedom from symptomatic AT/AF/AFL recurrence
Change in Blood interleukin-6 | 5 days pre-PFA and 48-72 hours post-PFA
  Inflammation is common among those with type 2 diabetes. Inflammatory markers (chemicals in the body that lead to inflammation), such as interleukin-6 (Il-6) have been found to be increased in those with type 2 diabetes
  For participants in substudy.
Change in C-reactive protein (CRP) | 5 days pre-PFA and 48-72 hours post-PFA
  C-reactive protein (CRP) is produced by the liver. The CRP test is a general test to check for inflammation in the body. It is not a specific test. This means it can reveal that inflammation somewhere in the body, but it cannot pinpoint the exact location or reason. The CRP test is often done with the ESR (erythrocyte or sedimentation rate) test which also looks for inflammation.
  For participants in substudy.
Changes in Tumor Necrosis Factor (TNF)-α | 5 days pre-PFA and 48-72 hours post-PFA
  Many people take medicines to reduce the immune system's abnormal response. These are called immunosuppressive medicines. Targeted drugs such as tumor necrosis factor (TNF) blockers can be used for some diseases.
  For participants in substudy.
Changes in Erythrocyte Sedimentation Rate (ESR) | 5 days pre-PFA and 48-72 hours post-PFA
  Erythrocyte sedimentation rate (ESR) is also commonly called a sed rate. It is a test that indirectly measures the level of certain proteins in the blood. This measurement correlates with the amount of inflammation in the body.
  For participants in substudy.
Brain natriuretic peptide (BNP) levels | 5 days pre-PFA and 48-72 hours post-PFA
  Brain natriuretic peptide (BNP) test is a blood test that measures levels of a protein called BNP that is made by the heart and blood vessels. BNP levels go up when the heart cannot pump the way it should. A result greater than 100 pg/mL is abnormal. The higher the number, the more likely heart failure is present and the more severe it is.
  For participants in substudy.
Change in durability of lesion sets in any patient that undergoes a second procedure | baseline (index procedure) and end of study 12 months
  Change in Durability of lesion sets in any patient that undergoes a second procedure (block across attempted lines, absence of electrograms in targeted substrate). Observe if the block(s) achieved at the targeted sites from the index procedure have persisted

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — The Mount Sinai Hospital, Icahn School of Medicine
Locations (5):
- United States (5):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Naples Comprehensive Health, Naples, Florida
  - The Mount Sinai Hospital, New York, New York
  - UPMC Pinnacle Hospitals, Harrisburg, Pennsylvania
  - Trident Medical Center, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Reddy VY, Anter E, Rackauskas G, Peichl P, Koruth JS, Petru J, Funasako M, Minami K, Natale A, Jais P, Nakagawa H, Marinskis G, Aidietis A, Kautzner J, Neuzil P. Lattice-Tip Focal Ablation Catheter That Toggles Between Radiofrequency and Pulsed Field Energy to Treat Atrial Fibrillation: A First-in-Human Trial. Circ Arrhythm Electrophysiol. 2020 Jun;13(6):e008718. doi: 10.1161/CIRCEP.120.008718. Epub 2020 May 8. PMID 32383391
- [Background] Reddy VY, Gerstenfeld EP, Natale A, Whang W, Cuoco FA, Patel C, Mountantonakis SE, Gibson DN, Harding JD, Ellis CR, Ellenbogen KA, DeLurgio DB, Osorio J, Achyutha AB, Schneider CW, Mugglin AS, Albrecht EM, Stein KM, Lehmann JW, Mansour M; ADVENT Investigators. Pulsed Field or Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2023 Nov 2;389(18):1660-1671. doi: 10.1056/NEJMoa2307291. Epub 2023 Aug 27. PMID 37634148
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Turagam MK, Neuzil P, Schmidt B, Reichlin T, Neven K, Metzner A, Hansen J, Blaauw Y, Maury P, Arentz T, Sommer P, Anic A, Anselme F, Boveda S, Deneke T, Willems S, van der Voort P, Tilz R, Funasako M, Scherr D, Wakili R, Steven D, Kautzner J, Vijgen J, Jais P, Petru J, Chun J, Roten L, Futing A, Lemoine MD, Ruwald M, Mulder BA, Rollin A, Lehrmann H, Fink T, Jurisic Z, Chaumont C, Adelino R, Nentwich K, Gunawardene M, Ouss A, Heeger CH, Manninger M, Bohnen JE, Sultan A, Peichl P, Koopman P, Derval N, Kueffer T, Rahe G, Reddy VY. Safety and Effectiveness of Pulsed Field Ablation to Treat Atrial Fibrillation: One-Year Outcomes From the MANIFEST-PF Registry. Circulation. 2023 Jul 4;148(1):35-46. doi: 10.1161/CIRCULATIONAHA.123.064959. Epub 2023 May 18. PMID 37199171
- [Background] Schmidt B, Bordignon S, Neven K, Reichlin T, Blaauw Y, Hansen J, Adelino R, Ouss A, Futing A, Roten L, Mulder BA, Ruwald MH, Mene R, van der Voort P, Reinsch N, Kueffer T, Boveda S, Albrecht EM, Schneider CW, Chun KRJ. EUropean real-world outcomes with Pulsed field ablatiOn in patients with symptomatic atRIAl fibrillation: lessons from the multi-centre EU-PORIA registry. Europace. 2023 Jul 4;25(7):euad185. doi: 10.1093/europace/euad185. PMID 37379528
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916